CLINICAL TRIAL: NCT07201467
Title: Phase 1b Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of KN060 in Patients With End Stage Renal Disease Receiving Regular Hemodialysis
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of KN060 in ESRD Dialysis Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KN060-C-102
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN060 (Experimental): KN060 diluted in normal saline and administered via proximal (arterial) dialysis line
  Interventions: Drug: KN060

INTERVENTIONS:
Drug: KN060 — pharmacokinetic and pharmacodynamic characteristics of KN060 in ESRD on Hemodialysis

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of KN060 in patients with end-stage renal disease on regular hemodialysis.

The secondary objectives to evaluate the pharmacokinetic and pharmacodynamic properties of multiple doses of KN060; to evaluate the immunogenicity of KN060; and to explore the efficacy of KN060 in preventing dialyzer and extracorporeal circuit thrombosis, arteriovenous fistula thrombosis in patients with end-stage renal disease undergoing regular hemodialysis. The main questions it aims to answer are:

* Whether KN060 is safe for ESRD dialysis patients
* Pharmacokinetic characteristics of KN060 in ESRD dialysis patients
* Whether KN060 can effectively prevent dialyzer and extracorporeal circuit thrombosis Researchers will evaluate the safety, tolerability, Pharmacokinetics and Pharmacodynamics profile, dialyzer and extracorporeal circuit thrombosis, arteriovenous fistula thrombosis of KN060 in ESRD dialysis patients

Subjects will :

* Eligible subjects will receive KN060 2.5 mg/kg every two weeks for a total of 6 doses.
* Assessed for the number, incidence, and severity of AEs, dialyzer thrombus, extracorporeal circuit thrombus, arteriovenous fistula thrombus, and time to hemostasis at the arteriovenous fistula puncture site.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 80 years (inclusive);
2. 1 8 kg /m ^2 <BMI <2 8 kg /m^2 ;
3. Diagnosis of ESRD and be receiving regular, stable hemodialysis treatment within the three months prior to screening: dialysis is performed through a functional, non-infected graft arteriovenous fistula / autologous arteriovenous fistula ( AVG/AVF ) ; dialysis is performed three times per week, with at least 3.5 hours per session ( at least 75% of dialysis sessions within the four weeks prior to randomization meet the this criteria) ;
4. The clinical status of the underlying ESRD is stable (assessed by the investigator) ;
5. Kt/V ≥ 1.2 within 3 months before screening ;
6. Male subjects: From the time they sign the informed consent form until 3 months after the last dose of KN060 , they agree to take effective contraceptive measures and avoid sperm donation ( effective contraceptive methods include: consistent scientific use of condoms , vasectomy , or partners who have undergone tubal ligation or hysterectomy, or have an intrauterine device implanted, etc. );
7. Women who are infertile and have no plans to have children (surgical infertility: such as after hysterectomy, bilateral salpingectomy , bilateral oophorectomy; or natural menopause: amenorrhea for ≥ 12 months and serum follicle-stimulating hormone (FSH) at menopausal levels ).

Exclusion Criteria:

1. A history of malignant tumor;
2. History of mechanical/artificial heart valve replacement surgery;
3. History of major medical events within 3 months before screening , such as acute coronary syndrome, stroke , major organ bleeding, acute heart failure, systemic thromboembolic events , major surgery, etc. , or history of AVF/AVG functional loss;
4. Using anticoagulant/antiplatelet drugs due to disease treatment , such as warfarin , dabigatran, rivaroxaban , clopidogrel , or aspirin >100 mg/day (investigators are allowed to use heparin / low molecular weight heparin during dialysis, depending on the situation );
5. There is a high risk of bleeding, or abnormal bleeding-related indicators:

1） Bleeding requiring hospitalization or clinically significant active bleeding within 3 months before screening ; prolonged arteriovenous fistula compression time within the past month; 2） Platelet count (PLT) <100 × 10^ 9 /L ( PLT between 75-100 × 10^9 /L , determined by the investigator after comprehensive evaluation), hemoglobin ( Hb ) < 90 g/L ; 3） Normalized ratio INR>1.4 , activated partial thromboplastin time ( APTT ) > 1.2 times ULN ; 4） Liver disease-related laboratory abnormalities: increased bleeding risk due to coagulation disorders , alanine aminotransferase (ALT) > 3 times ULN , aspartate aminotransferase ( AST) > 3 times ULN , total bilirubin (TB) > 2 times ULN and direct bilirubin proportion > 20%; 5） Poor blood pressure control in the past month before screening (judged by the investigator, such as repeated diastolic blood pressure ≥100 mmHg and/or systolic blood pressure ≥180 mmHg ) ; 6） Underwent brain, spinal or eye surgery (excluding cataract surgery) within three months before screening; 7） The patient has a bleeding disorder, a medical history that may increase the risk of bleeding, any condition that the investigator believes increases the risk of bleeding, or a history of severe bleeding disorders, such as massive gastrointestinal bleeding or cerebral hemorrhage ; 6. Supine blood pressure is < 90/50 mmHg , or > 170/100 mmHg (one retest is allowed) during screening; 7. Electrocardiogram during screening: heart rate < 45 beats / min or > 110 beats / min, QTcF > 500 ms, any significant arrhythmia or conduction abnormality ( e.g. Second degree or above atrioventricular block, preexcitation syndrome (except those who have undergone radical radiofrequency ablation) , non-sustained or sustained ventricular tachycardia (one retest is allowed); 8. History (<1 year) of drug or alcohol abuse or dependence before screening; 9. Have a history of allergy, or be allergic to the experimental drug/similar drugs or excipients; 10. Human immunodeficiency virus (HIV ) infection, syphilis infection, active HBV infection (HBV -DNA>ULN ), active HCV infection (HCV - RNA > ULN ) ; 11. Participated in another clinical trial and received trial drugs within 3 months before screening (signing ICF); 12. Plan to receive a kidney transplant during the trial or within 3 months after completing this trial; 13. Xanthine, coffee (small amounts of caffeine from normal food sources, such as chocolate, are permitted), or alcohol cannot be prohibited during the study; 14. Any concomitant disease or condition that the investigator believes may interfere with the study drug, affect study data, or pose a risk to patient safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety Results | up to 18 weeks
  Number, frequency, incidence and severity of treatment-emergent adverse events (TEAEs), drug-related adverse events (TRAEs), adverse events of special interest (AESIs), serious adverse events (SAEs), etc.

SECONDARY OUTCOMES:
Pharmacokinetics characteristics | up to 18 weeks
  Trough blood concentration after reaching stability (C min,ss )
Pharmacodynamic characteristics | up to 18 weeks
  Pharmacodynamic characteristics after multiple administrations, pharmacodynamic indicators include: total coagulation factor XI ( Total FXI ), free FXI ( Free FXI ), activated partial thromboplastin time ( APTT ) and FXI activity; After the blood drug concentration reached a stable level, the occurrence of achieving >50% or 95% inhibition of FXI;
Immunogenicity Results | up to 18 weeks
  The number and ratio of patients who produced anti-KN060 antibodies (ADA); the number and ratio of patients who produced anti-KN060 neutralizing antibodies (NAb) (NAb testing will be performed only on ADA-positive samples)
Bleeding Events | up to 18 weeks
  Number, frequency, and incidence of major bleeding events, clinically relevant non-major bleeding (CRNM) events, and all bleeding events;
Thrombosis events | up to 18 weeks
  Number, frequency, incidence and severity of dialyzer and extracorporeal circuit thrombosis, and arteriovenous fistula thrombosis
Time to hemostasis | up to 18 weeks
  Time to hemostasis at the arteriovenous fistula puncture site

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, Doctor, Principal Investigator — Peking University People's Hospital; Yuqing Chen, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No